CLINICAL TRIAL: NCT03446157
Title: Phase II Single-arm Study of the Combination of Palbociclib and Cetuximab in KRAS/NRAS/BRAF Wild-type Metastatic Colorectal Cancer
Brief Title: Palbociclib and Cetuximab in Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1717
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cancer of the Colon; Colon Cancer; Colon Neoplasms; Colonic Cancer; Neoplasms, Colonic
Keywords: colon cancer; metastatic colon cancer; palbociclib; cetuximab
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab; palbociclib

STUDY DESIGN:
Intervention Model Description: This is a multicenter, single-arm, phase II clinical trial of combination therapy with cetuximab and palbociclib in refractory KRAS, NRAS, and BRAF wild-type metastatic colorectal cancer (CRC) patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, single arm, Phase II (Experimental): Cetuximab and palbociclib
  Interventions: Drug: Cetuximab; Drug: Palbociclib

INTERVENTIONS:
Drug: Cetuximab — Loading dose on day 1 of week 1 of 400 mg/m2 via IV over 2 hours Subsequent doses of 250 mg/m2 via IV over 1 hour weekly for 4 weeks (28 days) in combination with palbociclib
  Other Names: Erbitux
Drug: Palbociclib — 125 mg taken orally once daily on days 1-21, then 7 days off
  Other Names: Ibrance

SUMMARY:
This research study is designed to provide a better understanding of study drugs cetuximab (Erbitux®) and palbociclib when used in combination to treat patients with metastatic colon cancer.

DETAILED DESCRIPTION:
This research study is designed to provide a better understanding of study drugs cetuximab (Erbitux®) and palbociclib when used in combination to treat patients with metastatic colon cancer.

Cetuximab (Erbitux®) is an antibody designed to target a protein called Epidermal Growth Factor Receptor (EGFR). EGFR plays an important role in the growth and survival of colon cancer. Antibodies are proteins that are naturally produced by the immune system and circulate throughout your body to help protect you from disease caused by bacteria, viruses, cancer cells or any foreign or toxic substance. Antibodies work by sticking to and flagging or marking foreign cells or substances so that your body's immune defense system will recognize, attack and remove them. Antibodies help the body rid itself of disease. Antibodies can also be designed in the laboratory to stick to specific parts of cancer cells (or normal cells) to change or block the ways those cells function in your body and to produce a therapeutic anti-cancer effect. Cetuximab (Erbitux®) is an antibody drug approved by the FDA and is commonly used to treat your type of colon cancer.

Palbociclib is an FDA-approved drug for patients with breast cancer. Palbociclib is not FDA-approved for the treatment of colon cancer, and is considered an investigational drug in this research study. Palbociclib targets a protein called CDK4/6 that is a critical part of the cell division and cell growth processes known as "the cell cycle". Laboratory studies have shown that palbociclib inhibits the cell cycle, slows or stops cell growth, and can cause cell death in cancer cells.

The combination of Cetuximab (Erbitux®) with palbociclib is not approved by the FDA for treating colon cancer and is considered investigational in this research study.

You are being asked to be in the study because your colon cancer has been found to contain the proteins KRAS, NRAS and BRAF that are normal (wild-type). These proteins play an important role in the growth and survival of colon cancer. This requirement is important because colon cancer with these characteristics has been shown to be more responsive to EGFR inhibitors such as cetuximab (Erbitux®), one of the drugs used in this study that is also a standard treatment option for your type of cancer. Also, Epidermal Growth Factor Receptor (EGFR) has been shown to stimulate cancer cell division, growth and survival by working together with KRAS, NRAS and BRAF to activate CDK4/6 and to support an accelerated cell cycle. This accelerated cell cycle allows the cancer cells to divide and grow faster than your normal cells but also can make them sensitive to the effects of CDK4/6 inhibitor palbociclib, a cell-cycle inhibitor.

To participate in this study you also must meet one of the following requirements:

A. You have not been treated with EGFR inhibitors such as cetuximab (Erbitux®) or panitumumab (Vectibix®).

B. You were treated with anti-EGFR drugs such as cetuximab (Erbitux®) or panitumumab (Vectibix®) and experienced at least 4 months of response to treatment, and it has been at least 8-weeks since you were last treated with an anti-EGFR drug.

This will allow investigators to compare the anti-cancer effects of cetuximab (Erbitux®) combined with palbociclib in 2 different groups of cancer patients:

1. Patients that have never received EGFR inhibitors like cetuximab (Erbitux®) or panitumumab (Vectibix®). This group will test whether resistance to the combination of cetuximab (Erbitux®) plus palbociclib develops in this type of cancer.
2. Patients that have previously shown an anti-cancer response to EGFR inhibitors, such as cetuximab (Erbitux®) or panitumumab (Vectibix®), of four or more months, but then developed resistance. This group will test whether the combination of cetuximab (Erbitux®) plus palbociclib is more effective against this resistant type of cancer.

Furthermore, laboratory studies have shown that the combination of EGFR and CDK inhibitors provide a stronger anti-cancer effect when used in combination than seen when each inhibitor is used alone. Thus, the reason researchers are using cetuximab (Erbitux®) and palbociclib in combination is to simultaneously target and inhibit multiple processes inside of the cancer cell that are critical to growth and survival of the tumor. With this combination strategy, researchers hope to improve upon existing anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

4.1.1 Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.

4.1.2 Age ≥ 18 years at the time of consent.

4.1.3 ECOG Performance Status of 0-2

4.1.4 Histologically-confirmed metastatic CRC

4.1.5 Measurable disease according to RECIST v1.1 for solid tumors.

4.1.6 Documented wild-type in KRAS and NRAS (codons 12, 13, 59, 61, 117, and 146) and in BRAF codon 600, based on tumor tissue taken from primary or metastatic site and tested for biomarkers

4.1.7 Previously treated with at least two prior regimens of systemic chemotherapy for metastatic or locally advanced, unresectable disease, including fluoropyrimidines (5-fluorouracil and/or capecitabine), oxaliplatin, and irinotecan.

A maintenance regimen of 5-fluorouracil or capecitabine, with or without bevacizumab, should not be counted as a separate line of treatment For patients who experienced disease recurrence during or within 6 months of completion of adjuvant chemotherapy with fluoropyrimidine and oxaliplatin, only one regimen of systemic chemotherapy for metastatic disease is required

4.1.8 Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained prior to initiating study medications.

System Laboratory Value Hematological* Hemoglobin (Hgb) ≥ 9 g/dL Absolute Neutrophil Count (ANC) ≥ 1500/mm3 Platelets ≥ 100,000/mm3

Renal* Creatinine OR Calculated creatinine clearance ≤1.5 x ULN

* 60 mL/min by Cockcroft-Gault formula Hepatic* Bilirubin ≤ 1.0 × upper limit of normal (ULN) Aspartate aminotransferase (AST) ≤ 3 × ULN OR

  * 5 × ULN (if liver metastases present) Alanine aminotransferase (ALT) ≤ 3 × ULN OR
  * 5 × ULN (if liver metastases present)

    * Note: Hematology and other lab parameters that are ≤ grade 2 BUT still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered adverse events unless they meet criteria for dose modification(s) of study medication outlined by the protocol and/or worsen from baseline during therapy.

4.1.9 Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to initiating study medications. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.

4.1.10 Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 6 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label.

4.1.11 Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 6 months after the last dose of study therapy.

4.1.12 Subjects is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

4.1.13 Able to swallow capsules, with no surgical or anatomic condition that will preclude the patient from swallowing and absorbing oral medications.

4.1.14 Has not undergone any major surgical procedures for at least 4 weeks, with full healing of all surgical wounds

4.1.15 At sites in the Southeastern U.S., subject must have negative serum test for galactose-alpha-1,3-galactose IgE See Appendix 12.5 for map (Note: positive test result is predictive of immediate-onset anaphylaxis reaction during first exposure to cetuximab, which is prevalent predominantly in limited geographic region of the Southeastern U.S. (Clin Mol Allergy 2012;10:1-11).

4.1.16 For Study Cohort A, has not had prior treatment with cetuximab, panitumumab, or other anti-EGFR therapy.

4.1.17 For Study Cohort B, must have had previous treatment with cetuximab or panitumumab with disease control (defined as complete response, partial response, or stable disease) lasting for ≥ 4 months in duration and completed their last anti-EGFR therapy 8 weeks prior to initiating treatment.

-

Exclusion Criteria:

4.2.1 Active infection requiring systemic therapy.

4.2.2 Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).

4.2.3 Presence of known, active central nervous system (CNS) metastases.

4.2.4 Treatment with any investigational drug within 28 days prior to initiating study medications.

4.2.5 Prior treatment with drug targeting cyclin-dependent kinase (CDK) family.

4.2.6 Subject is receiving prohibited medications or treatments as listed in section 5.5 of the protocol that cannot be discontinued/replaced by an alternative therapy.

4.2.7 Known hypersensitivity to the components of study drugs or analogs of study drugs.

4.2.8 Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.

4.2.9 Uncontrolled, severe concomitant comorbidity (e.g. uncontrolled hypertension, uncontrolled diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection).

4.2.10 History of interstitial lung disease or pneumonitis.

4.2.11 Any other clinically significant heart disease, including angina pectoris, resting bradycardia, left bundle branch block, ventricular tachyarrhythmia, unstable atrial fibrillation, acute myocardial infarction, or heart disease requiring cardiac pacemaker or implantable cardioverter/defibrillator

4.2.12 Known psychiatric or substance abuse disorder that would interfere with the ability of the patient to comply with trial requirements.

4.2.13 History of long-QT syndrome.

4.2.14 Baseline QTcF ≥ 470 msec.

4.2.15 Concomitant use of drugs known to cause QT prolongation as defined in Appendix 12.4 and in section 5.5 (Note: Ondansetron at doses ≤ 16 mg or less is allowed)

4.2.16 History of any of the following cardiovascular conditions within the past 6 months:

* Class III or IV congestive heart failure as defined by the New York Heart Association Criteria
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Symptomatic peripheral vascular disease or other clinically significant cardiac disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2026-01-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sanoff, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Sorah JD, Moore DT, Reilley MJ, Salem ME, Triglianos T, McRee AJ, Lee MS, Sanoff HK, Somasundaram AS. Phase II single-arm study of palbociclib and cetuximab in anti-EGFR naive patients with KRAS/NRAS/BRAF wild-type, metastatic colorectal cancer. Oncologist. 2025 Oct 1;30(10):oyaf305. doi: 10.1093/oncolo/oyaf305. PMID 40990835
- [Derived] Sorah JD, Moore DT, Reilley MJ, Salem ME, Triglianos T, Sanoff HK, McRee AJ, Lee MS. Phase II Single-Arm Study of Palbociclib and Cetuximab Rechallenge in Patients with KRAS/NRAS/BRAF Wild-Type Colorectal Cancer. Oncologist. 2022 Dec 9;27(12):1006-e930. doi: 10.1093/oncolo/oyac222. PMID 36288238
- [Derived] Noh JY, Lee IP, Han NR, Kim M, Min YK, Lee SY, Yun SH, Kim SI, Park T, Chung H, Park D, Lee CH. Additive Effect of CD73 Inhibitor in Colorectal Cancer Treatment With CDK4/6 Inhibitor Through Regulation of PD-L1. Cell Mol Gastroenterol Hepatol. 2022;14(4):769-788. doi: 10.1016/j.jcmgh.2022.07.005. Epub 2022 Jul 15. PMID 35843546
- See also: UNC Lineberger — http://unclineberger.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study between 03/23/2018 and 1/26/2023, at five cancer centers in the United States.
Pre-assignment Details: A total of thirty-three participants consented to the study, but nine of them were deemed to be ineligible and therefore were not enrolled in the study.
Groups:
- Cohort A: Subjects never received EGFR therapy.
- Cohort B: Subjects previously received EGFR therapy.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 13 | 11
Completed | 0 | 0
Not Completed | 13 | 11
Not completed — Death | 11 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Overall Response Rate (ORR) = CR + PR Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed assessed by Positron Emission Tomography (PET)- Computerized tomography (CT) scans. If the subject experienced a Complete Response (CR), the disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion new lesion.
Time Frame: 4 months
Population: Subjects started the study treatment and tumor response was assessed.1 subject was not included because they withdrew before starting the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 11
Participants
  Disease control (CR+PR+SD) achieved | 5 | 1
  Progression | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: as for outcome 1
Time Frame: 4 months (Cycle 5)
Population: Six subjects started the study treatment and tumor response was assessed were included in the analysis. The remaining 18 subjects were not included because they withdrew or did not survive.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 5 | 1
Participants
  Participants achieved (ORR) = CR + PR | 3 | 0
  Participants did not achieve (ORR) = CR + PR | 2 | 1

3. Secondary Outcome: Length of Overall Survival
Description: Time from the first day of treatment until death from any cause. All subjects who started the study treatment died or withdrew at 20 months.
Time Frame: Up to 20 months
Population: All subjects who started the study treatment were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 11
months | 13.9 [3.8 to 20] | 6.6 [1.4 to 9.6]

4. Secondary Outcome: Length of Progression Free Survival
Description: Time from the first day of treatment until disease progression as defined by RECIST or death from any cause.
  RECIST: Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  All subjects who started the study treatment died or withdrew at 20 months.
Time Frame: Up to 20 months
Population: Subjects started the study treatment and one subject was not included because they withdrew before starting the treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 11
months | 5.3 [2.7 to 8.8] | 1.8 [0.5 to 1.9]

5. Secondary Outcome: Number of Participants With Grade 3 and Grade 4 Adverse Events
Description: The number of participants who experienced treatment-related grade 3 and 4 toxicities defined by the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03) criteria.
  NCI CTCAE can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
  All subjects who started the study treatment died or withdrew at 20 months.
Time Frame: From day 1 of treatment until grade 3 or 4 events occurred. (Up to 20 monts)
Population: Subjects who started the study treatment Adverse Events were assessed.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Subjects did not receive EGFR Therapy previously f
- Cohort B: Subjects received EGFR Therapy previously
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 11
Participants
  Alkaline phosphatase increased | 0 | 1
  Anemia | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Fatigue | 0 | 1
  Hypocalcemia | 0 | 1
  Hypomagnesemia | 1 | 1
  Lymphocyte count decreased | 4 | 3
  Neutrophil count decreased | 2 | 1
  Platelet count decreased | 0 | 1
  Urticaria | 0 | 1
  Vomiting | 0 | 1
  White blood cell decreased | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the first day of study drug administration until 30 days after the completion of the last treatment (up to 20 months). Data on all-cause mortality were collected for up to 20 months.
Description: Any hospital admission was graded as a serious adverse event per protocol.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 11/13 | 9/11
Serious Adverse Events (participants affected / at risk) | 4/13 | 3/11
Other Adverse Events (participants affected / at risk) | 12/13 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=13) | Cohort B (N=11)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
fatigue (General disorders) | 0 | 1
fever (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
proteinuria (Renal and urinary disorders) | 0 | 1
Abdominal pain (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=13) | Cohort B (N=11)
Anemia (Blood and lymphatic system disorders) | 6 | 5
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 5
Hypothyroidism (Endocrine disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Watering eyes (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
vomiting (Gastrointestinal disorders) | 3 | 2
chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 2 | 0
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 1 | 1
Flu like symptoms (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 5 | 0
Pain (General disorders) | 4 | 0
Paronychia (Infections and infestations) | 0 | 1
Lung infection (General disorders) | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2
Alkaline phosphatase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 7 | 4
Blood bilirubin increased (Investigations) | 2 | 1
Creatinine increased (Investigations) | 4 | 1
Lymphocyte count decreased (Investigations) | 8 | 8
Neutrophil count decreased (Investigations) | 4 | 7
Platelet count decreased (Investigations) | 4 | 5
Weight loss (Investigations) | 3 | 0
White blood cell decreased (Investigations) | 6 | 8
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia (Investigations) | 1 | 2
Hypermagnesemia (Investigations) | 1 | 6
Hypoalbuminemia (Investigations) | 2 | 4
Hypocalcemia (Investigations) | 2 | 3
Hypokalemia (Investigations) | 1 | 4
Hypomagnesemia (Investigations) | 7 | 6
Hyponatremia (Investigations) | 3 | 1
Hypophosphatemia (Investigations) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 3 | 1
Hyperkalemia (Investigations) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 0
flank pain (General disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03446157/Prot_SAP_000.pdf